CLINICAL TRIAL: NCT03945019
Title: A Randomized, Placebo-Controlled, Double-Blind, Phase 3 Study to Evaluate the Efficacy and Safety of the Subcutaneous Injection of CT-P13 (CT-P13 SC) as Maintenance Therapy in Patients With Moderately to Severely Active Crohn's Disease
Brief Title: CT-P13 (Infliximab) Subcutaneous Administration in Patients With Moderately to Severely Active Crohn's Disease (LIBERTY-CD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P13 3.8; 2019-001087-30 (EudraCT Number)
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Results first posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-09

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CT-P13 SC (Experimental)
  Interventions: Biological: CT-P13 SC (Infliximab)
- Placebo SC (Placebo Comparator)
  Interventions: Other: Placebo SC

INTERVENTIONS:
Biological: CT-P13 SC (Infliximab) — Subcutaneous injection of CT-P13 SC
  Arms: CT-P13 SC
Other: Placebo SC — Subcutaneous injection of Placebo SC
  Arms: Placebo SC

SUMMARY:
This is Phase 3, Randomized, Placebo-controlled study to demonstrate superiority of CT-P13 SC over Placebo SC in Patients With Moderately to Severely Active Crohn's Disease

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female aged 18 to 75 years, inclusive.
* Patient who has moderately to severely active CD with a score on the CDAI of 220 to 450 points

Exclusion Criteria:

* Patient who has previously received either a TNFα inhibitor or biological agent within 5 half-lives
* Patient who has previously demonstrated inadequate response or intolerance to TNFα inhibitors for the treatment of CD.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2023-08-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- Biopharma Informatic - Houston, Houston, Texas, United States
- Vitebsk Regional Clinical Hospital, Vitebsk, Belarus
- Diagnostic and Consulting Center Aleksandrovska EOOD, Sofia, Bulgaria
- Clinical Hospital Centre Osijek, Osijek, Croatia
- Fakultni nemocnice Ostrava, Ostrava, Czechia
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France
- Praxis Prof. Herbert Kellner, München, Germany
- University General Hospital of Heraklion, Heraklion, Greece
- Debreceni Egyetem Klinikai Kozpont, Debrecen, Hungary
- Nirmal Hospital, Surat, India
- Sheba Medical Center, Ramat Gan, Israel
- Fondazione Policlinico Universitario A Gemelli-Rome, Roma, Italy
- Tsujinaka Hospital, Kashiwa, Japan
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- BRCR Global Mexico, Guadalajara, Mexico
- IMSP Institute of Clinical Cardiology, Chisinau, Moldova
- Hospital Nacional Cayetano Heredia, San Martín de Porres, Peru
- Poland (2):
  - Szpital Uniwersytecki Nr 2 im. dr Jana Biziela w Bydgoszczy, Centrum Endoskopii Zabiegowej, Poradnia, Bydgoszcz
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
- Dr.Carol Davila Emergency University Central Military Hospital, Bucharest, Romania
- Russia (2):
  - Klinika YZI 4D, Pyatigorsk
  - BioTekhServis, Saint Petersburg
- Clinical Hospital Centar Zvezdara, Belgrade, Serbia
- Fakultna nemocnica s poliklinikou F. D. Roosevelta, Banská Bystrica, Slovakia
- CLINRESCO, ARWYP Medical Suites, Johannesburg, South Africa
- Hospital Arquitecto Marcide, Ferrol, Spain
- Ege University Medical Faculty, Izmir, Turkey (Türkiye)
- Ukraine (2):
  - Communal Non-Commercial Enterprise Cherkasy Regional Hospital of Cherkasy Regional Council, Cherkassy
  - Municipal Nonprofit Enterprise Zaporizhzhia Regional Clinical Hospital Zaporizhzhia Regional Council, Zaporizhzhia

REFERENCES:
- [Derived] Colombel JF, Sandborn WJ, Schreiber S, Danese S, Klopocka M, Kierkus J, Kulynych R, Gonciarz M, Soltysiak A, Smolinski P, Sreckovic S, Valuyskikh E, Lahat A, Horynski M, Gasbarrini A, Osipenko M, Borzan V, Kowalski M, Saenko D, Sardinov R, Lee SJ, Kim S, Bae Y, Lee S, Lee S, Lee JH, Kim JM, Park G, Lee J, Lee J, Ryu JY, Sands BE, Hanauer SB. Subcutaneous infliximab (CT-P13 SC) as maintenance therapy for Crohn's disease and ulcerative colitis: 2-year results from open-label extensions of two randomized controlled trials (LIBERTY). J Crohns Colitis. 2025 Jun 4;19(6):jjaf060. doi: 10.1093/ecco-jcc/jjaf060. PMID 40243842
- [Derived] Hanauer SB, Sands BE, Schreiber S, Danese S, Klopocka M, Kierkus J, Kulynych R, Gonciarz M, Soltysiak A, Smolinski P, Sreckovic S, Valuyskikh E, Lahat A, Horynski M, Gasbarrini A, Osipenko M, Borzan V, Kowalski M, Saenko D, Sardinov R, Lee SJ, Kim S, Bae Y, Lee S, Lee S, Lee JH, Yang S, Lee J, Lee J, Kim JM, Park G, Sandborn WJ, Colombel JF. Subcutaneous Infliximab (CT-P13 SC) as Maintenance Therapy for Inflammatory Bowel Disease: Two Randomized Phase 3 Trials (LIBERTY). Gastroenterology. 2024 Oct;167(5):919-933. doi: 10.1053/j.gastro.2024.05.006. Epub 2024 May 23. PMID 38788861

RESULTS

PARTICIPANT FLOW:
Groups:
- CT-P13 IV 5mg/kg: Induction phase: Patients who enrolled received induction doses of CT-P13 5mg/kg via intravenous (IV) infusion at Weeks 0, 2, and 6.
- CT-P13 SC 120 mg: Maintenance phase: Patients who were classified as CDAI-100 responder at Week 10 received CT-P13 120 mg subcutaneously every 2 weeks from Week 10 to Week 54.
  From Week 22, patients who initially responded but then lost response could increase the dose to CT-P13 SC 240 mg (double injection [2 shots] of CT-P13 SC 120 mg) every 2 weeks.
- Placebo: Maintenance phase: Patients who were classified as CDAI-100 responder at Week 10 received placebo-matching subcutaneously every 2 weeks from Week 10 to Week 54.
  From Week 22, patients who initially responded but then lost response could increase the dose to CT-P13 SC 240 mg (double injection [2 shots] of CT-P13 SC 120 mg) every 2 weeks.
Period: Induction Phase
Arm/Group | CT-P13 IV 5mg/kg | CT-P13 SC 120 mg | Placebo
Started | 396 | 0 | 0
Completed | 343 | 0 | 0
Not Completed | 53 | 0 | 0
Period: Maintenance Phase
Arm/Group | CT-P13 IV 5mg/kg | CT-P13 SC 120 mg | Placebo
Started | 0 | 231 | 112
Completed | 0 | 196 | 87
Not Completed | 0 | 35 | 25

BASELINE CHARACTERISTICS:
Population: All-randomized population
Groups:
- CT-P13 SC 120 mg: CT-P13 SC 120 mg
- Placebo: Placebo
- Total: Total of all reporting groups
Arm/Group | CT-P13 SC 120 mg | Placebo | Total
Number analyzed (Participants) | 231 | 112 | 343
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (12.53) | 32.3 (11.53) | 34.8 (12.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 43 | 140
  Male | 134 | 69 | 203
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 5 | 13
  Asian | 9 | 4 | 13
  Black or African American | 1 | 0 | 1
  White | 211 | 101 | 312
  Other | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  Belarus | 3 | 3 | 6
  Bulgaria | 6 | 0 | 6
  Croatia | 12 | 2 | 14
  Czechia | 7 | 6 | 13
  France | 2 | 0 | 2
  Germany | 2 | 1 | 3
  Greece | 2 | 0 | 2
  Hungary | 6 | 6 | 12
  India | 4 | 2 | 6
  Israel | 13 | 4 | 17
  Italy | 9 | 5 | 14
  Japan | 3 | 2 | 5
  Latvia | 3 | 0 | 3
  Mexico | 8 | 5 | 13
  Moldova | 1 | 0 | 1
  Peru | 2 | 2 | 4
  Poland | 52 | 33 | 85
  Romania | 2 | 0 | 2
  Russia | 49 | 15 | 64
  Serbia | 6 | 7 | 13
  Slovakia | 1 | 4 | 5
  South Africa | 1 | 2 | 3
  Spain | 3 | 0 | 3
  Turkey | 1 | 0 | 1
  Ukraine | 29 | 13 | 42
  United States | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving Clinical Remission (Based on CDAI) at Week 54
Description: Clinical remission was defined as an absolute Crohn's Disease Activity Index (CDAI) score of <150 points.
  The total CDAI scores range from 0 to over 600 with higher scores indicating increased severity of disease. The index is the sum of 8 components; number of liquid or very soft stools, abdominal pain, general well-being, CD complications, taking antidiarrheal drugs, abdominal mass, hematocrit, and weight.
  Patients with dose adjustment to CT-P13 SC 240 mg prior to Week 54 were considered as non-remitter.
Time Frame: Week 54
Population: All-randomized population
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 SC 120 mg | Placebo
Number analyzed (Participants) | 231 | 112
Participants | 144 | 36
Statistical Analysis 1: Comparison: CT-P13 SC 120 mg vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by Previous biologic agent and/or JAK inhibitors exposure, Use of oral corticosteroids treatment at Week 0, Clinical remission at Week 10

2. Primary Outcome: Percentage of Patients Achieving Endoscopic Response (Based on Central SES-CD) at Week 54
Description: Endoscopic response was defined as a 50% decrease in Simplified Endoscopic Activity Score for Crohn's Disease (SES-CD) score from the baseline value.
  The SES-CD assesses the size of mucosal ulcers, ulcerated surface, endoscopic extension and the presence of stenosis. Each item is scored from 0-3, with total score from 0-60. Higher score indicates more severe endoscopic activity.
  Patients with dose adjustment to CT-P13 SC 240 mg prior to Week 54 were considered as non-responder.
  Statistical testing for this outcome based on the colonoscopy (SES-CD) was conducted using the colonoscopy reading results of central level.
Time Frame: Week 54
Population: All-randomized population
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 SC 120 mg | Placebo
Number analyzed (Participants) | 231 | 112
Participants | 118 | 20
Statistical Analysis 1: Comparison: CT-P13 SC 120 mg vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Patients Achieving CDAI-100 Response at Week 54
Description: Crohn's Disease Activity Index (CDAI)-100 response was defined as a decrease in CDAI score of 100 points or more from the baseline value.
  The total CDAI scores range from 0 to over 600 with higher scores indicating increased severity of disease. The index is the sum of 8 components; number of liquid or very soft stools, abdominal pain, general well-being, CD complications, taking antidiarrheal drugs, abdominal mass, hematocrit, and weight.
  Patients with dose adjustment to CT-P13 SC 240 mg prior to Week 54 were considered as non-responder.
Time Frame: Week 54
Population: All-randomized population
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 SC 120 mg | Placebo
Number analyzed (Participants) | 231 | 112
Participants | 152 | 43

4. Secondary Outcome: Percentage of Patients Achieving Clinical Remission (Based on AP and SF) at Week 54
Description: Clinical remission was defined as an average worst daily Abdominal Pain (AP) score of ≤1 (using 4-point scale) and an average daily loose/watery Stool Frequency (SF) score of ≤3 (of Type 6 or Type 7 on Bristol Stool Form Scale (BSFS)) with no worsening in either average score compared with the baseline value.
  AP score is patient recorded score on a scale 0 to 3 (none, mild, moderate, or severe) and higher score indicates severe abdominal pain. SF score is patient recorded number of loose/watery stool defined as BSFS type 6 or 7 per day. BSFS is an ordinal scale of stool types ranging from the hardest (Type 1) to the softest (Type 7).
  Patients with dose adjustment to CT-P13 SC 240 mg prior to Week 54 were considered as non-remitter.
Time Frame: Week 54
Population: All-randomized population
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 SC 120 mg | Placebo
Number analyzed (Participants) | 231 | 112
Participants | 131 | 35

5. Secondary Outcome: Percentage of Patients Achieving Endoscopic Remission (Based on Central SES-CD) at Week 54
Description: Endoscopic remission was defined as an absolute Simplified Endoscopic Activity Score for Crohn's Disease (SES-CD) score of ≤4 and at least 2-point reduction from the baseline value with no segment sub-score of >1.
  The SES-CD assesses the size of mucosal ulcers, ulcerated surface, endoscopic extension and the presence of stenosis. Each item is scored from 0-3, with total score from 0-60. Higher score indicates more severe endoscopic activity.
  Patients with dose adjustment to CT-P13 SC 240 mg prior to Week 54 were considered as non-remitter.
Time Frame: Week 54
Population: All-randomized population
Measure: Count of Participants; unit: Participants
Groups:
- Placebo SC: Placebo
Arm/Group | CT-P13 SC 120 mg | Placebo SC
Number analyzed (Participants) | 231 | 112
Participants | 80 | 12

ADVERSE EVENTS:
Time Frame: For CT-P13 SC and Placebo groups, the overall summary of Treatment-Emergent Adverse Events during the maintenance period (from Week 10 to Week 54) was reported. For CT-P13 IV 5mg/kg group, the overall summary of Treatment-Emergent Adverse Events during the induction phase (from Week 0 to prior to Week 10, before initiation of CT-P13 SC administeration) was reported.
Description: Safety analyses were pre-specified to only report the most severe event if the same events were occurred to the same patient.
  For CT-P13 IV 5mg/kg group, the safety analyses were performed ITT population. For CT-P13 SC and Placebo groups, the safety analyses were performed in the safety population. Analysis of safety population were performed based on the actual treatment group and differences from the randomized population accordingly.
Groups:
- CT-P13 IV 5 mg/kg: Patients who administered CT-P13 IV 5mg/kg at Week 0, 2, and 6.
- CT-P13 SC 120 mg (Including 240 mg): Patients who administered CT-P13 SC 120 mg every 2 weeks from W10 to Week 54. Patients who received adjusted dose of CT-P13 SC 240mg which is allowed from Week 22 are also included.
- CT-P13 SC 120 mg: Patients who administered CT-P13 SC 120 mg every 2 weeks from W10 to Week 54. For patients who received adjusted dose of CT-P13 SC 240mg, data collected before initiation of dose adjustment are included.
- CT-P13 SC 120 mg to 240 mg: Patients who administered CT-P13 SC 120 mg every 2 weeks from W10 and initiated adjusted dose of CT-P13 SC 240mg which is allowed from Week 22.
- Placebo: Patients who administered Placebo every 2 weeks from W10 to Week 54. For patients who received adjusted dose of CT-P13 SC 240mg, data collected before initiation of dose adjustment are included.
Arm/Group | CT-P13 IV 5 mg/kg | CT-P13 SC 120 mg (Including 240 mg) | CT-P13 SC 120 mg | CT-P13 SC 120 mg to 240 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/396 | 1/238 | 1/238 | 0/45 | 0/105
Serious Adverse Events (participants affected / at risk) | 12/396 | 16/238 | 15/238 | 1/45 | 8/105
Other Adverse Events (participants affected / at risk) | 51/396 | 75/238 | 70/238 | 9/45 | 30/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P13 IV 5 mg/kg (N=396) | CT-P13 SC 120 mg (Including 240 mg) (N=238) | CT-P13 SC 120 mg (N=238) | CT-P13 SC 120 mg to 240 mg (N=45) | Placebo (N=105)
Anaemia (study drug unrelated) (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Cardiovascular insufficiency (study drug unrelated) (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Crohn's disease (study drug unrelated) (Gastrointestinal disorders) | 6 | 3 | 3 | 0 | 1
Haemorrhoids (study drug unrelated) (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Intestinal obstruction (study drug unrelated) (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Intestinal perforation (study drug unrelated) (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Subileus (study drug unrelated) (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Accidental death (study drug unrelated) (General disorders) | 0 | 1 | 1 | 0 | 0
Abdominal abscess (study drug unrelated) (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Abdominal sepsis (study drug unrelated) (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Abdominal wall abscess (study drug unrelated) (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Abscess intestinal (study drug unrelated) (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Anal abscess (study drug unrelated) (Infections and infestations) | 1 | 1 | 1 | 0 | 0
Appendicitis (study drug unrelated) (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Arthritis bacterial (study drug related) (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Bartholinitis (study drug unrelated) (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Bronchiolitis (study drug unrelated) (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Cytomegalovirus colitis (study drug related) (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Intestinal tuberculosis (study drug related) (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Orchitis (study drug unrelated) (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Peritonitis (study drug unrelated) (Infections and infestations) | 2 | 0 | 0 | 0 | 1
Urinary tract infection (study drug related) (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Humerus fracture (study drug unrelated) (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Infusion related reaction (study drug related) (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Skin laceration (study drug unrelated) (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Blood creatine phosphokinase increased (study drug related) (Investigations) | 0 | 0 | 0 | 0 | 1
Intervertebral disc degeneration (study drug unrelated) (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Colon cancer stage III (study drug unrelated) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Altered state of consciousness (study drug unrelated) (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Neurovascular conflict (study drug unrelated) (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Mixed anxiety and depressive disorder (study drug unrelated) (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Psychotic disorder (study drug unrelated) (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (study drug unrelated) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (study drug unrelated) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Acne fulminans (study drug unrelated) (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P13 IV 5 mg/kg (N=396) | CT-P13 SC 120 mg (Including 240 mg) (N=238) | CT-P13 SC 120 mg (N=238) | CT-P13 SC 120 mg to 240 mg (N=45) | Placebo (N=105)
Anaemia (Blood and lymphatic system disorders) | 16 | 13 | 11 | 3 | 5
Crohn's disease (Gastrointestinal disorders) | 10 | 12 | 11 | 1 | 17
Injection site reaction (General disorders) | 2 | 14 | 11 | 3 | 1
COVID-19 (Infections and infestations) | 10 | 27 | 22 | 5 | 5
Headache (Nervous system disorders) | 18 | 18 | 18 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT03945019/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/19/NCT03945019/SAP_001.pdf